CLINICAL TRIAL: NCT01184534
Title: Increasing Patient Preparedness for the Procedural Experience and Improving Qualitative Outcomes Through Patient Education
Brief Title: Multimedia Patient Education
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-0397
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: Lung Biopsy; Multimedia patient education tool; Multimedia Education Tool; Computed tomography guided lung biopsy; Computerized Tomography; CT; Questionnaire; Lung nodules
MeSH Terms: conditions — Lung Neoplasms | interventions — Videotape Recording; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Questionnaires + Video
  Interventions: Behavioral: Video
- Questionnaires
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Video — 5 minute multimedia presentation (video)
  Groups: Questionnaires + Video
Behavioral: Questionnaires — 2 questionnaires pre and post procedure taking approximately 15 minutes each to complete.
  Other Names: Survey
  Groups: Questionnaires

SUMMARY:
Objective:

To compare changes in patient anxiety levels between groups of patients who either were or were not exposed to an informative multimedia patient education tool, in order to determine how the addition of such a multimedia tool will affect this parameter. Specifically, the study will focus on subjective anxiety as measured on pre procedure and post procedure patient surveys as detailed under study components.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will complete a questionnaire that asks how you feel before the procedure. It will take about 5 minutes to complete.

After you have completed the questionnaire, you will be randomly assigned (as in the flip of a coin) to Group 1 or Group 2. You will have an equal chance of being in either group.

If you are in Group 1, you will receive routine information before the lung biopsy and you will watch a video on a handheld or laptop machine with headphones. The video is designed to help you understand the biopsy procedure. This video should last about 5 minutes. You will then complete a questionnaire that asks how you feel after watching the video. It will take about 5 minutes to complete.

If you are in Group 2, you will receive routine information before the lung biopsy. You will then complete another questionnaire that asks how you feel before the procedure. It will take about 5 minutes to complete.

After your routine lung biopsy, both groups will complete a questionnaire that asks how you feel after the procedure. It will take about 5 minutes to complete.

For Group 1, the total time to complete the questionnaires and watch the video will be 20 minutes.

For Group 2, the total time to complete the questionnaires will be 15 minutes.

Length of Study:

Your participation in this study will be over once you complete the questionnaire after your lung biopsy.

This is an investigational study.

Up to 100 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for a computed tomography (CT) guided lung biopsy
2. Literate English-speaking

Exclusion Criteria:

1. Refusal to participate
2. Current diagnosis of psychosis, dementia or other mentally altered state.
3. Monitored anesthesia care (MAC) or general endotracheal anesthesia (GETA) during the procedure.
4. Patients who are clinically diagnosed as hearing and visually impaired.
5. Patients who have had prior image guided biopsies in our department.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UT MD Anderson Cancer Center Patients scheduled for a computed tomography (CT) guided lung biopsy
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Patient Response to Subjective Anxiety Surveys | 1 day (pre and post lung biopsy procedure)
  Subjective anxiety as measured on pre procedure and post procedure patient surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen McRae, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org